CLINICAL TRIAL: NCT00896935
Title: Arizona Cancer Center Biospecimen Repository
Status: Recruiting | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000597579; P30CA023074 (NIH); UARIZ-06-0609-04 (Other: University of Arizona); UARIZ-BIO#A06035 (Other: University of Arizona); UARIZ-SRC18042 (Other: University of Arizona)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tissue will be collected and preserved from the primary organ site, from the metastases, from patient blood (serum and lymphocytes), from patient urine, and from related samples of other tissues/fluids removed by the surgeon left over after diagnostic testing.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: biologic sample preservation procedure — biologic sample preservation procedure

SUMMARY:
RATIONALE: Collecting and storing samples of tissue and blood from patients with cancer to test in the laboratory may help the study of cancer in the future.

PURPOSE: This research study is collecting and storing tumor, tissue, and blood samples from patients with pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide cancer investigators access to a wide variety of tissues and biospecimens for translational studies in cancer.
* Collect and preserve tissue from the primary organ site (uninvolved and involved with cancer), from the metastases, from patient blood (serum and lymphocytes), and from patient urine.
* Provide quality-controlled storage and management of the specimen bank.
* Collect relevant clinical and pathologic information with appropriate privacy protection.
* Contribute to the development of a comprehensive database annotated with relevant clinical data, pathology, and research findings.

OUTLINE: This is a multicenter study.

Tumor samples, lymph node samples, and normal pancreas tissue samples are collected. Blood samples are also collected prior to surgery, six months after the initial blood draw and tissue sample collection, and every six months thereafter for two years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient who is seen at the Arizona Cancer Center or University Medical Center and will undergo any surgery or procedure for cancer

PATIENT CHARACTERISTICS:

* NA

PRIOR CONCURRENT THERAPY:

* NA

As this is a biospecimen repository, participation is open to all cancer patients being treated at the Arizona Cancer Center or University Medical Center by investigators on this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The goal of this protocol is to provide cancer investigators access to a wide variety of tissues and biospecimens for translational studies in cancer by collecting and preserving tissue from the primary organ site, from the metastases, from patient blood (serum and lymphocytes), from patient urine, and from related samples of other tissues/fluids removed by the surgeon left over after diagnostic testing. No additional tissue will be taken at the time of surgery other than that required for patient care, but additional blood and urine samples will be obtained at that time. This protocol is not limited to certain types of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2006-08-01 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Provision of tissue samples and biospecimens for translational study | July 2024
  An electronic record of the specimens is kept in a secure, web-based database. Follow-up information from patients will be obtained from the patient medical record, and updated every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Setsuko K. Chambers, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/publications/pdq